CLINICAL TRIAL: NCT01208506
Title: First Human Dose Trial of NNC0114-0000-0005 in Healthy Subjects and Subjects With Rheumatoid Arthritis
Brief Title: First-in-Man Trial of NNC114-0005 in Healthy Subjects and Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NN8828-3837; 2010-018347-33 (EudraCT Number); U1111-1116-2585 (Other: WHO)
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Inflammation; Rheumatoid Arthritis; Healthy
MeSH Terms: conditions — Inflammation; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Dose level 1 (Experimental)
  Interventions: Drug: NNC0114-0000-0005; Drug: placebo
- Dose level 2 (Experimental)
  Interventions: Drug: NNC0114-0000-0005; Drug: placebo
- Dose level 3 (Experimental)
  Interventions: Drug: NNC0114-0000-0005; Drug: placebo
- Dose level 4 (Experimental)
  Interventions: Drug: NNC0114-0000-0005; Drug: placebo
- Dose level 5 (Experimental)
  Interventions: Drug: NNC0114-0000-0005; Drug: placebo
- Dose level 6 (Experimental)
  Interventions: Drug: NNC0114-0000-0005; Drug: placebo
- Dose level 7 (Experimental)
  Interventions: Drug: NNC0114-0000-0005; Drug: placebo
- Dose level 8 (Experimental)
  Interventions: Drug: NNC0114-0000-0005; Drug: placebo

INTERVENTIONS:
Drug: NNC0114-0000-0005 — A single dose of NNC0114-0000-0005 administered i.v. (into the vein) in healthy subjects.
  Arms: Dose level 1; Dose level 2; Dose level 3; Dose level 7
Drug: NNC0114-0000-0005 — A single dose of NNC0114-0000-0005 administered i.v. (into the vein) in healthy subjects. Based on safety data, a single dose of NNC0114-0000-0005 may be administered i.v. (into the vein) in subjects with RA. In addition a single dose of NNC0114-0000-0005 administered s.c. (under the skin) in healthy subjects.
  Arms: Dose level 4
Drug: NNC0114-0000-0005 — A single dose of NNC0114-0000-0005 administered i.v. (into the vein) in healthy subjects. In addition a single dose of NNC0114-0000-0005 may be administered s.c. (under the skin) in healthy subjects based on safety data.
  Arms: Dose level 5
Drug: NNC0114-0000-0005 — A single dose of NNC0114-0000-0005 administered i.v. (into the vein) in healthy subjects. Based on safety data, a single dose of NNC0114-0000-0005 may be administered i.v. (into the vein) in subjects with RA. In addition a single dose of NNC0114-0000-0005 may be administered s.c. (under the skin) in healthy subjects based on safety data.
  Arms: Dose level 6
Drug: NNC0114-0000-0005 — A single dose of NNC0114-0000-0005 administered i.v. (into the vein) in healthy subjects. Based on safety data, a single dose of NNC0114-0000-0005 may be administered i.v. (into the vein) in subjects with RA.
  Arms: Dose level 8
Drug: placebo — A single dose of NNC0114-0000-0005 placebo.

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the safety, tolerability, pharmacokinetic (the effect of the body on the investigated drug), pharmacodynamic biomarkers (biomarkers related to anti-IL-21 expected mode of action) and signs of clinical efficacy of increasing single doses, at 9 i.v. (into the vein) dose levels in Healthy Subjects , at 3 i.v. dose levels in subjects with rheumatoid arthritis (RA) and at 3 s.c. dose levels in Healthy Subjects.

ELIGIBILITY:
Inclusion Criteria:

* For all subjects the following applies:
* Male subjects, if not sterilized, must be using two acceptable methods of contraception (e.g., spermicidal gel plus condom) for the entire duration of the trial corresponding to up to three months following trial drug administration. Male subjects must also agree to refrain from sperm donation from screening (trial start) until 120 days beyond trial drug administration
* For healthy subjects (HS) the following additional criteria applies:
* Male subjects, aged between 18 and 60 years (both inclusive) and in good health, as determined by past medical history, physical examination, vital signs, (electrocardiogram) ECG, and laboratory tests at screening (trial start)
* For subjects with rheumatoid arthritis (RA) the following additional criteria applies:
* Diagnosed with RA at least 3 months prior to trial drug administration
* Active RA, characterised by a Disease Activity Score 28 (DAS28)-C-reactive protein (CRP) greater than 3.2
* Effective methods of contraception
* Male and female subjects aged greater and equal to 18 and greater and equal to 75 years
* Females must be post-menopausal or surgically sterile (post-menopausal for at least 1 year). If female of child-bearing potential must be willing to use highly effective method of birth control during the trial until their final visit
* Methotrexate treatment (MTX) treatment for at least 12 weeks at a stable dose (dose at least 7.5 mg/week and maximum 25 mg/week inclusive) for at least 4 weeks prior to trial product administration
* Concomitant medication according to specific list

Exclusion Criteria:

* For all subjects the following applies:
* Body mass index (BMI) between 20.0-38.0 kg/m2 (both inclusive)
* Females with a positive pregnancy test
* History of regular alcohol consumption exceeding 14 drinks per week for females or 21 drinks per week for men
* Donation or loss of at least 400 mL of blood within 8 weeks prior to trial product administration
* For healthy subjects (HS) the following additional criteria applies:
* Body weight greater than 110.0 kg
* For subjects with rheumatoid arthritis (RA) the following additional criteria applies:
* Chronic inflammatory autoimmune disease other than RA (except secondary Sjögren's syndrome or stable hypothyroidism)
* History of or current inflammatory joint disease other than RA such as gout (crystal proven), psoriatic arthritis, juvenile idiopathic arthritis, current reactive arthritis or Lyme disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | at least 12 weeks after dose administration

SECONDARY OUTCOMES:
Area under the serum concentration-time curve | at least 12 weeks after dose administration
Maximum level of free IL-21 and maximum level of bound IL-21 in peripheral blood | at least 12 weeks after dose administration
Change in Disease Activity Score 28 (DAS28)-C-reactive protein (CRP) in subjects with RA | at least 12 weeks after dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

REFERENCES:
- [Result] First in human study with recombinant anti-IL-21 monoclonal antibody in healthy subjects and patients with rheumatoid arthritis. Arthritis and Rheumatism 2012; 64 (10 (supplement)): Abstract 1279
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com